CLINICAL TRIAL: NCT04758624
Title: Elucidating the Temporality of Structural and Functional Connectivity Changes in Essential Tremor After Successful Deep Brain Stimulation to the Dentato-rubro-thalamic Tract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-20-0739
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
Keywords: deep brain stimulation
MeSH Terms: conditions — Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Deep Brain Stimulation(DBS) (Experimental)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Medtronic Activa device will be implanted and administered clinically, except as part of the trial after 24 months of DBS being on it will be turned off for 3 days and will be turned back on.

SUMMARY:
The purpose of this study is to elucidate the structural connectivity of the dentato-rubro-thalamic tract (DRTt) and to detect functional network changes due to DRTt stimulation

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of Essential Tremor, made by a movement disorder neurologist, where tremor is not secondary to any disease process or traumatic insult
* distal appendicular tremor, with minimal proximal component
* tremor refractory to multiple medication regimens and/or where the medications cause intolerable side effects
* tremor judged to be severely impacting their quality of life.

Exclusion Criteria:

* significant neurological disorder
* significant dementia or neurocognitive limitations as assessed by neuropsychiatry (when necessary)
* severe psychiatric illness with suicidal ideations
* previous surgery to destroy the target region of the brain
* surgical contraindications to DBS
* current major medical problems that affect brain anatomy,neurochemistry, or function, e.g., liver insufficiency, kidney insufficiency, cardiovascular problems, systemic infections, cancer, hypothyroidism, auto-immune diseases, and any current of history of brain disorder (seizure disorder, stroke, dementia, meningitis, encephalitis, degenerative neurologic diseases and head injury with loss of consciousness for any period of time)
* family history of hereditary neurologic disorder, besides essential tremors ET
* floating metallic objects in the body
* pregnancy
* alcohol or substance abuse/dependence in the past 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Structural connectivity as indicated by fractional anisotropy (FA) as measured by diffusion tensor imaging (DTI) MRI | Baseline before DBS implant
Structural connectivity as indicated by fractional anisotropy (FA) as measured by diffusion tensor imaging (DTI) MRI | 24 months after start of DBS
Structural connectivity as indicated by mean diffusivity as measured by diffusion tensor imaging (DTI) MRI | Baseline before DBS implant
Structural connectivity as indicated by mean diffusivity as measured by diffusion tensor imaging (DTI) MRI | 24 months after start of DBS
Structural connectivity as indicated by radial diffusivity as measured by diffusion tensor imaging (DTI) MRI | Baseline before DBS implant
Structural connectivity as indicated by radial diffusivity as measured by diffusion tensor imaging (DTI) MRI | 24 months after start of DBS
Structural connectivity as indicated by axial diffusivity as measured by diffusion tensor imaging (DTI) MRI | Baseline before DBS implant
Structural connectivity as indicated by axial diffusivity as measured by diffusion tensor imaging (DTI) MRI | 24 months after start of DBS
Functional connectivity as indicated by blood oxygen level dependent (BOLD) signal as measured by resting state functional MRI (rsfMRI) | Baseline before DBS implant
Functional connectivity as indicated by blood oxygen level dependent (BOLD) signal as measured by resting state functional MRI (rsfMRI) | 24 months after start of DBS
Functional connectivity as indicated by blood oxygen level dependent (BOLD) signal as measured by resting state functional MRI (rsfMRI) | Baseline before DBS is turned off
Functional connectivity as indicated by blood oxygen level dependent (BOLD) signal as measured by resting state functional MRI (rsfMRI) | 72 hours after DBS is turned off
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | Baseline before DBS implant
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | 24 months after start of DBS
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | Baseline before DBS is turned off
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | 72 hours after DBS is turned off
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | During DBS placement surgery before active DBS
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Tremor as assessed by score on The Essential Tremor Rating Scale (TETRAS) | During DBS placement surgery during active DBS
  10 items are measured-each is scored from 0-4,higher number indicating more tremor
Spectral power recorded during intraoperative electrocorticography (ECoG) | During DBS placement surgery before active DBS
Spectral power recorded during intraoperative electrocorticography (ECoG) | During DBS placement surgery during active DBS

SECONDARY OUTCOMES:
Ataxia as assessed by score on the Scale for the Assessment and Rating of Ataxia (SARA) | Baseline before DBS implant
  It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Ataxia as assessed by score on the Scale for the Assessment and Rating of Ataxia (SARA) | 24 months after start of DBS
  It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Ataxia as assessed by score on the Scale for the Assessment and Rating of Ataxia (SARA) | Baseline before DBS is turned off
  It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Ataxia as assessed by score on the Scale for the Assessment and Rating of Ataxia (SARA) | 72 hours after DBS is turned off
  It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Tremor amplitude as assessed by accelerometric power | Baseline before DBS is turned off
Tremor amplitude as assessed by accelerometric power | 72 hours after DBS is turned off

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Fenoy, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conner CR, Forseth KJ, Lozano AM, Ritter R 3rd, Fenoy AJ. Thalamo-cortical evoked potentials during stimulation of the dentato-rubro-thalamic tract demonstrate synaptic filtering. Neurotherapeutics. 2024 Jan;21(1):e00295. doi: 10.1016/j.neurot.2023.10.005. Epub 2023 Dec 19. PMID 38237402